CLINICAL TRIAL: NCT06991153
Title: Impact of Lung Boost Device on Ventilatory Functions and Fatigue in Patients With Interstitial Lung Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Mokhtar Mahmoud Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005083
Record Dates: First submitted 2024-12-03; First posted 2025-05-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Interstitial Lung Disease
MeSH Terms: conditions — Lung Diseases, Interstitial | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lung Boost Device Training + Traditional physical therapy program + Medical Treatment (Experimental): Twenty patients will receive respiratory training using lung boost 3 sessions per week for 8 weeks plus maintain their medical treatment.
  Interventions: Device: Lung Boost Device Training; Other: Traditional physical therapy program; Drug: Medical Treatment
- Traditional physical therapy program + Medical Treatment (Active Comparator): Twenty patient will receive traditional physical therapy program in addition to medical treatment.
  Interventions: Other: Traditional physical therapy program; Drug: Medical Treatment

INTERVENTIONS:
Device: Lung Boost Device Training — Patients in the experimental group will train with the Lung Boost Respiratory Trainer (MD800) for 8 weeks, three times weekly, totaling 24 sessions. The procedure will be explained, and equipment sanitized before use. Training begins in strength mode at level 1, where patients inhale deeply through a mouthpiece, with feedback provided via on-screen balls. If level 5 is easily reached, resistance increases using a cone, restarting at level 1. Sessions include 15 repetitions of 2-3 second inhalations and exhalations, performed in three sets with 15-second rests to prevent fatigue. In endurance mode, patients inhale or exhale as long as possible, progressing gradually from level 1. Each session lasts 15 minutes, divided into three sets of five breaths with 15-second rests. This structured program enhances respiratory muscle strength and endurance.
  Arms: Lung Boost Device Training + Traditional physical therapy program + Medical Treatment
Other: Traditional physical therapy program — Patients in both groups will receive a traditional physical therapy program for the chest in form of diaphragmatic breathing exercise and pursed-lip breathing exercise for 8 weeks.
Drug: Medical Treatment — Patients in both groups will receive medical treatment for 8 weeks.
  Other Names: corticosteroids

SUMMARY:
The purpose of this study will be to determine the effect of lung boost exercise on ventilatory functions, fatigue, and physical function capacity in Interstitial lung disease patients.

DETAILED DESCRIPTION:
Death rates from chronic respiratory diseases have recently increased, largely driven by the rising burden of interstitial lung diseases (ILDs) doubling mortality rates over the past 4 decades. Pulmonary fibrosis (PF), a form of ILD, is characterized by destruction of lung tissue and accounts for the highest increase in mortality rates.

According to the Global Burden of Disease Study, between the years of 1990 and 2013, there was an 86% increase in ILD related years of life lost, and, for the first time, among the top 50 causes of global years of life lost.

In patients with ILD next to dyspnea, fatigue is expected to be the most prevalent symptom. Surprisingly, the prevalence of severe fatigue has been scarcely studied in ILD patients and limited information on its associated factors is available.

ILDs are associated with skeletal muscle dysfunction, worsening exercise capacity, and poor health-related quality of life.

So,This study will explore the impact of lung boost on ventilatory function, fatigue and physical function capacity in interstitial lung disease patients and may give a suggestion of therapeutic modality that is easy and applicable groups of patients to decrease the symptoms and improve the quality of life for this patients.

ELIGIBILITY:
Inclusion Criteria:

1. Forty female patients have Interstitial lung disease .
2. All patients diagnosed as ILD on clinical and radiological basis.
3. Age will range between 45 to 55 years old .
4. All patients will be with mild hypoxemia range from 90 to 92 oxygen saturation
5. They have Interstitial lung disease for at least 3 years ago.
6. Stable in medical and hemodynamic state

Exclusion Criteria:

1. Cardiovascular (as acute heart failure, unstable angina or recent myocardial infarction)
2. Patients with other significant respiratory disorders such as acute infections, pulmonary tuberculosis, chronic obstructive pulmonary disease, asthma, bronchiectasis, lung carcinoma, and pneumothorax.
3. cognitive impairments, history of cerebrovascular accident, active cancer will be excluded.
4. Hepatitis, cirrhosis.
5. Current treatment for cancer or active infection
6. Orthopedic problem.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-05-29 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
Forced vital capacity (FVC) | 8 weeks
  It will be assessed for all participants before and after treatment, using an electronic spirometer .
The first second of forced expiration (FEV1) | 8 weeks
  It will be assessed for all participants before and after treatment, using an electronic spirometer .
FEV1/FVC ratio | 8 weeks
  It will be assessed for all participants before and after treatment, using an electronic spirometer .
Fatigue Severity Scale (FSS) | 8 weeks
  It will be used to measure fatigue severity for all participants before and after treatment. The FSS is one of the most frequently used inventories for measuring fatigue in people with chronic illnesses. The original FSS is a nine-item questionnaire developed to measure fatigue severity as a unidimensional concept. Each FSS item consists of statements that are scored on a seven-point Likert type scale, ranging from 1 ("strongly disagree") to 7 ("strongly agree").

SECONDARY OUTCOMES:
oxygen saturation (SpO2) | 8 weeks
  It will be assessed for all participants before and after treatment, using a pulse oximetry, which is a simple, non-invasive, widely available medical tool that measures oxygen saturation (SpO2) through a device attached to a finger, a toe or an earlobe.
6-min walk test (6MWT) | 8 weeks
  It will be used to assess functional exercise capacity for all participants before and after treatment. The 6MWT is a validated tool, of submaximal intensity, Used to objectively measure functional exercise capacity. Individual walks without assistance for 6 minutes and the distance is measured.
King's Brief Interstitial Lung Disease (K-BILD) questionnaire | 8 weeks
  It will be used to assess health impairments induced by ILD for all participants before and after treatment. The questionnaire covers 15 questions spread out in three domains ("breathlessness and activity", "chest symptoms" and "psychological impact") via a seven point Likert Scale. The total (cross-domain) score and domain-specific subscores range from zero to 100 with higher values indicating better health.

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen Gharib El Nahas, PhD, Study Chair — Professor, Cairo university
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt